CLINICAL TRIAL: NCT02836587
Title: The Influence of Balance Training on Postural Control in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Zdenek Svoboda, Ph.D., Palacky University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UPOL_FTK_001
Record Dates: First submitted 2016-06-07; First posted 2016-07-19 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Accidental Falls

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- interventional (Experimental): Experimental group will undergo balance training for 8 weeks.
  Interventions: Behavioral: Balance training
- control (No Intervention): Control group will have no assigned intervention.

INTERVENTIONS:
Behavioral: Balance training — The interventional program will last 8 weeks with the intensity of two 60-minutes lectures a week. Training sessions will be delivered by a physiotherapist to small groups of patients (3-5). Participants will receive individualized exercises which will be focused on main 4 types - stance exercises, gait and transition exercises and strength exercises especially focused on muscle strength of the lower extremities. The difficulty level will be increased progressively after participant's ability to complete each exercise independently (e.g. eyes closed, exercises on balance equipment - wobble board, foam etc., addition of a secondary cognitive task). The training session will consist of a ten-minute warm-up followed by five-minute stretching, 30 minutes of balance training and 15 minutes of stretching and relaxation.
  Arms: interventional

SUMMARY:
Fall related injuries are major health problem which effect especially elderly population. After experiencing a fall, most of the elderly are unable to resume their previous mobility and the fear of future falls affects their daily life. Falls in elderly population are often related to balance or gait problems. The aim of this study is to assess the influence of balance training on postural and motor control of healthy elderly participants. The study is designed as a parallel interventional study with experimental and control group (allocation ratio 1:1). Participants' general health, balance abilities, fear of falling and gait stability and variability will be assessed on the baseline measurement, right after and 2 months after the completion of the training programme. Experimental group will undergo training focused on development of balance abilities and strength twice a week (60 minutes in length each) for 8 weeks. Participants will receive individualized exercises which will be focused on the main 4 types - stance exercises, gait and transition exercises and strength exercises especially focused on muscle strength of lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* age 60+
* ability to stand and walk without aid or support
* participation in the institutional program "Falls risk and balance assessment" with successful completion of one year of observation for falls

Exclusion Criteria:

* neuromuscular or orthopaedic impairments that severely limit mobility and balance
* surgery or injury on the musculoskeletal system less than 2 years before baseline measurement
* any acute illness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-16 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline Berg balance scale score after completing intervention | 2 months
Change from baseline mean velocity of centre of pressure during quiet stance after completing intervention | 2 months
Change from baseline stride time variability after completing intervention | 2 months

SECONDARY OUTCOMES:
Change from baseline Falls efficacy scale - International score after completing intervention | 2 months
Change from baseline gait velocity after completing intervention | 2 months
Change from baseline short-term Lyapunov exponents after completing intervention | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Zdenek Svoboda, Ph.D., Principal Investigator — Faculty of Physical Culture, Palacky University Olomouc
Locations (1):
- Faculty of Physical Culture, Palacky University Olomouc, Olomouc, Czechia